CLINICAL TRIAL: NCT01428310
Title: A Single Center, Single-Blind, Randomized, Crossover Pilot Study to Evaluate the Safety and Effects of Anatabloc™, a Dietary Supplement, in Reducing the Urge to Smoke in Daily Smokers Followed by an Open-Label Extension
Brief Title: Study to Evaluate the Safety and Efficacy of Dietary Supplement Anatabloc in Reducing Daily Smokers' Urge to Smoke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rock Creek Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: RCP-006
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Tobacco Use Disorder; Tobacco Dependence; Smoking
Keywords: dietary supplement; nutraceutical
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anatabloc(TM) (Active Comparator): dissolvable bit containing dietary ingredients, binders, fillers, and flavors
  Interventions: Dietary Supplement: Anatabloc(TM)
- CigRx(R) (Active Comparator): dissolvable bit containing dietary ingredients, binders, fillers, and flavors
  Interventions: Dietary Supplement: CigRx(R)

INTERVENTIONS:
Dietary Supplement: Anatabloc(TM) — one dissolvable bit, one time, after a period of abstinence from smoking
  Arms: Anatabloc(TM)
Dietary Supplement: CigRx(R) — one dissolvable bit, one time, after a period of abstinence from smoking
  Arms: CigRx(R)

SUMMARY:
This study will consist of 2 phases. Phase 1 will be a one day crossover study to see the effects of study product on a smoker's desire to smoke, measured by changes in scores on questionnaires given over time. Phase 2 will be a two-week extension, in which subjects will self-administer the study product and visit the study site for assessment of desire to smoke and collection of samples for the evaluation of smoking-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult smokers
* using at least 1 pack of cigarettes per day, for at least 5 years

Exclusion Criteria:

* allergy to study product components

Ages: 23 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
effect on subject's craving to smoke | 5 hours
  craving is assessed by changes in questionnaire answers over time

SECONDARY OUTCOMES:
adverse events related to study product | 5 hours
  collection of information on adverse events related to study product

CONTACTS AND LOCATIONS:
Overall Officials: Maria Varga, MD, Principal Investigator — Star Scientific, Inc
Locations (1):
- Comfort Inn, Martinsburg, West Virginia, United States